CLINICAL TRIAL: NCT04743518
Title: Impact of Anti-TNF, Vedolizumab and Tofacitinib on Aortic Stiffness, Carotid Intima-media Thickness and Cardiovascular Risk of Patients With Ulcerative Colitis
Acronym: VASC-UC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2020_843_0114
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis; cardiovascular risk; CIMT
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Carotid Intima-Media Thickness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- anti-TNF (Active Comparator)
  Interventions: Other: Aortic pulse wave velocity; Other: carotid intima media thickness (CIMT)
- vedolizumab (Active Comparator)
  Interventions: Other: Aortic pulse wave velocity; Other: carotid intima media thickness (CIMT)
- tofacitinib (Active Comparator)
  Interventions: Other: Aortic pulse wave velocity; Other: carotid intima media thickness (CIMT)

INTERVENTIONS:
Other: Aortic pulse wave velocity — Aortic pulse wave velocity (aPWV) is a measure of aortic stiffness
Other: carotid intima media thickness (CIMT) — carotid intima media thickness (CIMT)

SUMMARY:
An increased risk of cardiovascular (CV) diseases has been observed in patients with inflammatory bowel diseases (IBD). The impact of IBD drugs, such as anti-TNF, anti-integrins or anti-JAK, on the risk of CV events in IBD is remains unknown. Aortic pulse wave velocity (aPWV), a measure of aortic stiffness, and carotid intima media thickness (CIMT) are both predictors of cardiovascular events and are increased in patients with IBD. The investigators aimed to prospectively compare the CV risk, CIMT, arterial stiffness and biomarkers of endothelial dysfunction at baseline and after 3 and 12 months of anti-TNF, vedolizumab and tofacitinib.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis evolving for at least 6 months,
* Patient older than 18 years,
* Initiating a treatment by infliximab, adalimumab, golimumab, vedolizumab or tofacitinib,
* Written informed consent.

Exclusion Criteria:

* Patients with anti-hypertensive, antiplatelet or lipid-lowering drugs without stable dosage within the 3 months before the study and over the study period,
* Patients with a cardiovascular event such as myocardial infarction and stroke,
* Diabetic patient,
* Pregnant women,
* Minor
* people unable to give their consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
variation of carotid intima media thickness (CIMT) between the 3 patient groups | at the end of month 3

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No